CLINICAL TRIAL: NCT03251911
Title: An Open Label Study to Investigate the Role of Ivacaftor (VX-770) for the Treatment of Chronic Bronchitis With CFTR Dysfunction
Brief Title: VX-770 for the Treatment of Chronic Bronchitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, George Solomon, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F160914011
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Chronic Bronchitis
MeSH Terms: conditions — Bronchitis, Chronic | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivacaftor (VX770) (Experimental): Ivacaftor (VX-770) for the Treatment of Chronic Bronchitis with CFTR Dysfunction
  Interventions: Drug: Ivacaftor (VX-770)

INTERVENTIONS:
Drug: Ivacaftor (VX-770) — of Ivacaftor (VX-770) for the Treatment of Chronic Bronchitis with CFTR Dysfunction

SUMMARY:
This research study will test how well a new drug affects bronchiectasis or chronic bronchitis. The new drug, Ivacaftor (KALYDECO), is a drug that has recently been approved by the U.S. Food and Drug Administration (FDA) for patients with a lung disease called Cystic Fibrosis (CF). It has not been approved for use in patients with bronchiectasis or chronic bronchitis.

DETAILED DESCRIPTION:
The study is an open label study of orally-administered ivacaftor in subjects with chronic bronchitis and/or bronchiectasis. Subjects will be administered the study drug ivacaftor 150 mg twice daily (BID). The study drug is commercially available and will be purchased by the participant.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18 years
* A Clinical diagnosis of Bronchiectasis and/or Chronic Bronchitis in the investigators opinion
* Exhibit symptoms of chronic bronchitis as defined by the Medical Research Council
* FEV1 percent predicted greater than 40 percent Post Bronchodilator
* Clinically stable in the last 4 weeks with no evidence of exacerbation
* Weight of 40 kg to120 kg
* Willingness to use at least one form of acceptable birth control including abstinence, condom with spermicide, or hormonal contraceptives
* Willing to monitor blood glucose if known history of diabetes mellitus requiring insulin or medical therapy
* Element of CFTR Dysfunction, as defined by Sweat Chloride

Exclusion

* Daytime use of Oxygen Therapy
* Documented history of drug abuse within the last year
* Subjects should not have a pulmonary exacerbation or changes in therapy for pulmonary disease within 28 days before receiving the first dose of study drug.
* Cirrhosis or elevated liver transaminases > 3X ULN
* GFR < 50 estimated by Cockroft-Gault
* Any illness or abnormal lab finding that, in the opinion of the investigator might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Pregnant or Breastfeeding
* Subjects taking any inhibitors or inducers of CYP3A4, including certain herbal medications and grapefruit juice. (Excluded medications and foods including the drugs and foods are provided in the appendix document)
* Uncontrolled Diabetes
* Clinically significant arrhythmias or conduction abnormalities that in the opinion of the investigator that affect patient safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
change in lung function | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No